CLINICAL TRIAL: NCT01193478
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Escalating, Multiple, Oral Doses of GS 5885 in Treatment Naïve Subjects With Chronic Genotype 1 Hepatitis C Virus Infection
Brief Title: A Multiple Ascending Dose Study of GS 5885 in Previously Untreated Subjects With Genotype 1 Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-256-0102
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: HCV Infection
Keywords: Hepatitis C; HCV RNA; multiple ascending dose; NS5A; GS-5885; chronic genotype 1 HCV infection
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 (Active Comparator): GS-5885 (3 mg), once daily or matching placebo, once daily
  Interventions: Drug: GS-5885; Drug: Placebo
- Cohort 2 (Active Comparator): GS-5885 (10 mg), once daily or matching placebo, once daily
  Interventions: Drug: GS-5885; Drug: Placebo
- Cohort 3 (Active Comparator): GS-5885 (30 mg), once daily or matching placebo, once daily
  Interventions: Drug: GS-5885; Drug: Placebo
- Cohort 4 (Active Comparator): GS-5885 ( up to 90 mg), once daily or matching placebo, once daily
  Interventions: Drug: GS-5885; Drug: Placebo
- Cohort 5 (Active Comparator): GS-5885 (up to 90 mg), once daily or matching placebo, once daily
  Interventions: Drug: GS-5885; Drug: Placebo
- Cohort 6 (optional) (Active Comparator): GS-5885 (up to 90 mg), once daily or matching placebo, once daily
  Interventions: Drug: GS-5885; Drug: Placebo

INTERVENTIONS:
Drug: GS-5885 — tablet, oral, 3 mg once daily for 3 days
  Arms: Cohort 1
Drug: Placebo — tablet, oral, once daily for 3 days
  Arms: Cohort 1
Drug: GS-5885 — tablet, oral, 10 mg once daily for 3 days
  Arms: Cohort 2
Drug: Placebo — tablet, oral, once daily for 3 days
  Arms: Cohort 2
Drug: GS-5885 — tablet, oral, 30 mg once daily for 3 days
  Arms: Cohort 3
Drug: Placebo — tablet, oral, once daily for 3 days
  Arms: Cohort 3
Drug: GS-5885 — tablet, oral, up to 90 mg once daily for 3 days
  Arms: Cohort 4
Drug: Placebo — tablet, oral, once daily for 3 days
  Arms: Cohort 4
Drug: GS-5885 — tablet, oral, up to 90 mg once daily for 3 days
  Arms: Cohort 5
Drug: Placebo — tablet, oral, once daily for 3 days
  Arms: Cohort 5
Drug: GS-5885 — tablet, oral, up to 90 mg once daily for 3 days
  Arms: Cohort 6 (optional)
Drug: Placebo — tablet, oral, once daily for 3 days
  Arms: Cohort 6 (optional)

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and activity of escalating, multiple, oral doses of GS-5885 in subjects with chronic genotype 1 Hepatitis C Virus (HCV) infection. Each participant in the study will be sequestered in the clinic for the initial 5 days of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronically infected with HCV genotype 1
* HCV treatment-naïve
* Not co-infected with HIV or HBV
* HCV RNA viral load of at least 100,000 IU/mL
* BMI 19 to 35 kg/m2
* Subject agrees to use highly effective contraception methods if female of childbearing potential or sexually active male.

Exclusion Criteria:

* History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* Decompensated liver disease or cirrhosis or evidence of hepatocellular carcinoma
* Serological evidence of co-infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or another HCV genotype
* Subjects with known, current use of amphetamines and/or cocaine; subjects taking methadone or buprenorphine (opioid replacement therapy) or ongoing alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting an adverse event or experiencing a laboratory abnormality | Safety and tolerability assessments will be performed up to Study Day 14 following administration of multiple doses of GS-5885 or placebo for 3 days
Antiviral activity measures: measured by change in plasma HCV RNA levels form baseline | Assessed up to Study Day 14 following administration of multiple doses of GS-5885 or placebo for 3 days

SECONDARY OUTCOMES:
Measure of GS-5885 plasma concentration over time | Assessed up to Study Day 14 following administration of multiple doses of GS-5885 or placebo for 3 days
Emergence of viral resistance | Up to 48 weeks following Study Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Diana Brainard, MD, Study Director — Gilead Sciences
Locations (13):
- United States (13):
  - Anaheim, California
  - Cypress, California
  - National City, California
  - Washington D.C., District of Columbia
  - DeLand, Florida
  - Miami, Florida
  - Orlando, Florida
  - St Louis, Missouri
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
  - Tacoma, Washington

REFERENCES:
- [Derived] Wong KA, Worth A, Martin R, Svarovskaia E, Brainard DM, Lawitz E, Miller MD, Mo H. Characterization of Hepatitis C virus resistance from a multiple-dose clinical trial of the novel NS5A inhibitor GS-5885. Antimicrob Agents Chemother. 2013 Dec;57(12):6333-40. doi: 10.1128/AAC.02193-12. Epub 2013 Jul 22. PMID 23877691